CLINICAL TRIAL: NCT00076050
Title: Bone Sparing Effects of Soy Phytoestrogens in Menopause
Brief Title: Using Soy Estrogens to Prevent Bone Loss and Other Menopausal Symptoms
Acronym: SPARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Silvina Levis, MD, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AR048932 (NIH); R01AR048932 (NIH); NIAMS-114; SPARE
Record Dates: First submitted 2004-01-13; First posted 2004-01-14 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Menopause; Osteoporosis; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive a 200-mg dose of soy isoflavones daily over 2 years.
  Interventions: Dietary Supplement: Soy isoflavones
- 2 (Placebo Comparator): Participants will receive placebo daily over 2 years.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soy isoflavones — Purified soy isoflavones (phytoestrogens) in tablet form tablets; 200 mg.
  Arms: 1
Dietary Supplement: Placebo — Placebo soy isoflavones
  Arms: 2

SUMMARY:
The purpose of this study is to determine if soy-derived phytoestrogens (naturally occurring compounds similar to estrogen) can prevent bone loss and other menopausal symptoms in women who have recently gone through menopause.

Study hypothesis: Tablets of high-dose, purified soy phytoestrogens spare the normally occurring spinal bone loss and improve biological and other emotional changes of menopause.

DETAILED DESCRIPTION:
The risks of bone loss and osteoporosis increase significantly after menopause. Although hormone therapy (HT) can spare menopausal women from bone loss and other menopausal symptoms, Women's Health Initiative (WHI) findings indicate significant potential health risks associated with HT. This has prompted women to switch from HT to naturally occurring compounds similar to estrogen, such as those derived from soy, in the hope that estrogens from plant sources can provide benefits while sparing adverse effects caused by prescribed estrogens. However, the long-term efficacy and safety of plant estrogens are unknown. This study will evaluate the effectiveness of treatment using purified soy isoflavones, a dietary source of phytoestrogens, in preventing bone loss, menopausal symptoms, and other changes associated with estrogen deficiency in young menopausal women. The "Soy Phytoestrogens As Replacement Estrogen (SPARE)" study will provide a foundation of knowledge from which menopausal women and their doctors can begin to make more informed decisions regarding HT and other treatment options.

Enrollment into the study will occur over 3 years, with each participant taking part in the study for a total of 2 years. Participants will be randomly assigned to one of two groups; the first group will receive a 200 mg dose of soy isoflavones daily and the second group will receive placebo daily. There will be 10 study visits: screening, study entry, randomization at Month 1, six follow-up visits at Months 2, 4, 8, 12, 16, 20, and a final visit at the end of active participation at Month 24. At each study visit, participants will have blood drawn, provide urine samples, answer questionnaires, and have mammograms and bone density tests.

ELIGIBILITY:
Inclusion Criteria

* Absence of menstrual period for 12 months but not more than 5 years, or absence of menstrual period for 6 to 12 months and follicle stimulating factor (FSH) greater than 40 IU/L

Exclusion Criteria

* Treatment with estrogens, progesterone, raloxifene, or tamoxifen
* Treatment with bisphosphonates, calcitonin, fluoride, or systemic corticosteroids
* Use of soy/herbal supplements, including DHEA, within 3 months prior to study entry
* Use of antibiotics in the month prior to study entry
* Use of prescription medication to treat hot flashes
* Chemical menopause, including post-chemotherapy
* Hyperthyroidism
* Hypothyroidism
* Uncontrolled diabetes
* Malabsorption syndromes or other chronic diseases
* Body mass index (BMI) less than 20 or greater than 32
* Bone mineral density (BMD) T-score below -2.0 in lumbar spine or femoral neck

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2003-09; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvina Levis, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

REFERENCES:
- [Derived] Levis S, Strickman-Stein N, Ganjei-Azar P, Xu P, Doerge DR, Krischer J. Soy isoflavones in the prevention of menopausal bone loss and menopausal symptoms: a randomized, double-blind trial. Arch Intern Med. 2011 Aug 8;171(15):1363-9. doi: 10.1001/archinternmed.2011.330. PMID 21824950

RESULTS

PARTICIPANT FLOW:
Groups:
- Soy Isoflavone Group: A total of 122 participants were randomized to receive a 200-mg dose of soy isoflavones in tablet form daily by mouth, over 2 years. The medication was delivered in four tablets that had to be taken fasting in the morning.
- Placebo Group: A total of 126 participants were randomized to receive placebo tablets by mouth daily over 2 years.The medication was delivered in four tablets that had to be taken fasting in the morning.
Period: Overall Study
Arm/Group | Soy Isoflavone Group | Placebo Group
Started | 122 | 126
Completed | 99 | 83
Not Completed | 23 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Soy Isoflavone Group | Placebo Group | Total
Number analyzed (Participants) | 122 | 126 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 126 | 248
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (3.3) | 52 (3.3) | 52.5 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 126 | 248
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 122 | 126 | 248

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bone Mineral Density
Time Frame: baseline and 2 years
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Soy Isoflavone Group | Placebo Group
Number analyzed (Participants) | 99 | 83
g/cm2 | 1.146 (0.125) | 1.132 (0.124)

2. Secondary Outcome: Changes in Women's Health Questionnaire Score
Description: This self-administered questionnaire contains 23 items, distributed among 6 factors: anxiety and depressed mood (7 items), well-being (4 items), somatic symptoms (5 items), memory and concentration (3 items), vasomotor symptoms (2 items) and sleep problems (2 items). The instrument has a structured format and the response choices consist of 4-point Likert scales ('yes definitely' to 'no, not at all'). Item scores are collapsed into a dichotomous scale, where higher scores indicate a greater level of symptomatology or difficulty; i.e., if the response is 1 or 2 (positive response), the score = 1; if the response is 3 or 4 (negative response), the score is 0. Results can be reported as a total score, where the range is 0-23, but also for each dimension. Thus, the ranges of the subscales are: for anxiety and mood 0-7, for well-being 0-4, somatic symptoms 0-5, memory and concentration 0-3, vasomotor symptoms 0-2 and sleep problems 0-2.
Time Frame: baseline and 2 years
Measure: Mean (Standard Error); unit: change in score
Arm/Group | Soy Isoflavone Group | Placebo Group
Number analyzed (Participants) | 99 | 83
change in score | -0.73 (0.54) | -0.34 (0.77)

3. Secondary Outcome: Change in Vaginal Maturation Value
Description: The Vaginal Maturation Value (VMV) describes the proportion of the three vaginal epithelial cell types (parabasal, intermediate and superficial) obtained from a swab of the vaginal walls. The changes in the proportion of each type of cells reflects the degree of exposure to estrogen of the vaginal epithelium. The VMV lists the percentage of each type of cell appearing on the smear, with the total of all three values equaling 100%. The index is read from left to right; i.e. VMI of 5/40/55 represents 5% parabasal cells, 40% intermediate cells and 55% superficial cells. Exposure to estrogens results in some parabasal cells, a greater proportion of intermediate cells and few superficial cells.
Time Frame: baseline and 2 years
Measure: Mean (Standard Error); unit: score
Arm/Group | Soy Isoflavone Group | Placebo Group
Number analyzed (Participants) | 99 | 83
score | 0.20 (2.53) | -1.78 (2.86)

ADVERSE EVENTS:
Groups:
- Soy Isoflavones: A total of 122 participants were randomized to receive a 200-mg dose of soy isoflavones in tablet form daily by mouth, over 2 years. The medication was delivered in four tablets that had to be taken fasting in the morning.
- Placebo: A total of 126 participants were randomized to receive placebo tablets by mouth daily over 2 years.The medication was delivered in four tablets that had to be taken fasting in the morning.
Arm/Group | Soy Isoflavones | Placebo
Serious Adverse Events (participants affected / at risk) | 9/122 | 3/126
Other Adverse Events (participants affected / at risk) | 121/122 | 122/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soy Isoflavones (N=122) | Placebo (N=126)
fracture (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
breast cancer (Reproductive system and breast disorders) | 1 (1) | 1 (1)
leukemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soy Isoflavones (N=122) | Placebo (N=126)
abdominal bloating (Gastrointestinal disorders) | 64 | 54
headache (Nervous system disorders) | 54 | 43
hair loss (Skin and subcutaneous tissue disorders) | 39 | 43
dry mouth (Gastrointestinal disorders) | 35 | 37
constipation (Gastrointestinal disorders) | 38 | 26
breast tenderness (Reproductive system and breast disorders) | 31 | 30
edema of lower exteremity (Skin and subcutaneous tissue disorders) | 19 | 19
vaginal bleeding (Reproductive system and breast disorders) | 17 | 18
anorexia (Gastrointestinal disorders) | 21 | 12
abnormal mammogram (Reproductive system and breast disorders) | 9 | 6
joint tenderness (Musculoskeletal and connective tissue disorders) | 6 | 7
tenderness lower extremities (Musculoskeletal and connective tissue disorders) | 3 | 9
upper respiratory track infection (Respiratory, thoracic and mediastinal disorders) | 7 | 5
urinary track infection (Renal and urinary disorders) | 7 | 5
hypertension (Cardiac disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No